CLINICAL TRIAL: NCT03079492
Title: Magnetic Resonance Imaging of Neonates With Hypoxic Ischemic Encephalopathy Before and During Moderate Hypothermia
Brief Title: MRI of Neonate With HIE Before and During the Moderate Hypothermia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: 2016YFC0100300HIE01
Record Dates: First submitted 2017-03-08; First posted 2017-03-14 (Actual); Last update posted 2017-03-14 (Actual); Status verified 2017-02

CONDITIONS: Hypoxic-Ischemic Encephalopathy
MeSH Terms: conditions — Hypoxia-Ischemia, Brain | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Magnetic resonance imaging — Magnetic resonance imaging will be used to estimate brain temperature and cerebral blood flow

SUMMARY:
Moderate hypothermia has been demonstrated to be the effective treatment for neonates with hypoxic-ischemic encephalopathy (HIE). However, few studies reveal the actual alterations in physiological parameters (i.e. brain temperature and cerebral blood flow) of neonates undergoing cooling, especially for HIE lesions. Therefore, this project aims to utilize the magnetic resonance imaging (MRI), i.e. MR thermal imaging and phase contrast MRI to measure the changes of these parameters before and during hypothermia; and then make comparisons with the routine nasopharyngeal and rectal temperature. All these would provide in vivo quantitative data for therapeutic evaluation and promote the optimization.

DETAILED DESCRIPTION:
1. Study objects 1.1 Primary object To examine the changes of brain temperature and cerebral blood flow in neonates with HIE before and during (i.e. cooling lasting for 24~36 hr) selective brain cooling.

   1.2 Secondary object To compare the differences in temperature between brain (thalamus and HIE lesions) and nasopharynx and rectum of HIE neonates during the cooling.
2. Methods Prospective observational study; the MR thermal imaging and phase contrast MRI will be used to estimate brain temperature and cerebral blood flow.

Neonates with HIE who fulfilled the moderate hypothermia criteria will be recruited from the neonatal intensive care units. MR scans will be performed twice after informed parental consent. The first scan will be before the hypothermia and the second scan will be during the hypothermia. The first scan will be performed while the neonate is still in the intensive care unit. At the time of the second MR scan, the neonate is still in the intensive care unit, and the neonate in hypothermia group is receiving the brain selective cooling. Sedation would be used if required in these babies.

ELIGIBILITY:
Inclusion Criteria:

* Neonates in the neonatal intensive care unit who fulfill the hypothermia criteria for treating the hypoxic ischemic encephalopathy and who are scheduled to have an MRI for evaluation of the extent of their injury.
* Parents, clinicians and physician consent to perform evaluation of MRI before and during the hypothermia.

Exclusion Criteria:

* Neonates too unstable to have MRI exam, defined by being more than 40% oxygen on the ventilator.
* Hypothermia treatment interruption caused by potential factors.
* Neonates with central nervous system infection,intracranial hemorrhage and brain parenchyma lesions caused by trauma.

Ages: 6 Hours to 4 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates with hypoxic-ischemic encephalopathy who fulfill the moderate hypothermia criteria
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-06-01 (Estimated); Primary Completion 2019-05-31 (Estimated); Study Completion 2020-05-31 (Estimated)

PRIMARY OUTCOMES:
Cooling-induced changes in brain temperature and cerebral blood flow | before and during (cooling lasting for 24~36 hr) the hypothermia
  Magnetic resonance imaging will be used to measure the changes of brain temperature and cerebral blood flow before and during the brain selective cooling

CONTACTS AND LOCATIONS:
Overall Officials: Chao Jin, Phd, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- the First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, China

IPD SHARING:
Plan to Share IPD: No